CLINICAL TRIAL: NCT04962503
Title: A Proof of Concept, Phase IIa, Open Label Study to Evaluate the Safety of Afamelanotide in Patients With Acute Arterial Ischaemic Stroke (AIS) Due to Distal [M2 Segment and Beyond] Arterial Large Vessel Occlusion (LVO) or Perforator Occlusion and Who Are Ineligible for Intravenous Thrombolysis (IVT) or Endovascular Thrombectomy (EVT)
Brief Title: A Proof of Concept Study to Evaluate the Safety of Afamelanotide in Patients With Acute Arterial Ischaemic Stroke (AIS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Clinuvel Pharmaceuticals Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CUV801
Record Dates: First submitted 2021-06-23; First posted 2021-07-15 (Actual); Results first posted 2023-04-11 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-03

CONDITIONS: Arterial Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — afamelanotide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Afamelanotide (Experimental)
  Interventions: Drug: Afamelanotide

INTERVENTIONS:
Drug: Afamelanotide — Six adult patients with clots located in the higher segments of the brain and who are ineligible for alternative treatments will be enrolled in the study and evaluated for six weeks. The study will assess patients' brain injury with computed tomography (CT) scans and magnetic resonance imaging (MRI), as well as using recognised methods of clinical evaluation to measure changes in patients' neurological and cognitive function following treatment.

SUMMARY:
The primary study objective is to assess the safety of afamelanotide while the secondary objective is to assess whether the therapy affects the size of the penumbra, by increasing blood flow, restoring oxygen supply to the brain, and reducing the amount of cerebral oedema (fluid) which is seen as a result of the stroke. Positive findings would indicate that the drug is able to support brain tissue-at-risk and provide overall neuroprotection and benefit to stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects with a diagnosis of first AIS due to distal [M2 segment and beyond] occlusion or perforator occlusion
* Perfusion abnormalities observed on Computed Tomography Perfusion (CTP)
* Mild to moderate stroke severity
* Pre-stroke mRS <4
* Written informed consent obtained from patient and/or medical treatment decision maker prior to study-start (upon admission).

Exclusion Criteria:

* Administration of intravenous thrombolytic therapy in distal occlusion as etiology of AIS
* Intervention by endovascular thrombectomy (EVT)
* Known allergy or anaphylaxis to adrenocorticotropic hormone (ACTH) or melanocortins or any of the excipients listed in the Investigator's Brochure
* Any evidence of hepatic (defined as three times standard range) or renal impairment (defined as estimated glomerular filtration rate (eGFR) <50 mL/min/1.73 m²)
* Any other medical condition which may interfere with the study protocol
* Female who is pregnant (confirmed by positive serum beta human chorionic gonadotropin (β-HCG) pregnancy test prior to baseline) or lactating
* Females of child-bearing potential (pre-menopausal, not surgically sterile) not using adequate contraceptive measures (i.e. oral contraceptives, diaphragm plus spermicide, intrauterine device) or a lifestyle excluding pregnancy
* Unable to undergo MRI brain evaluation
* Not suitable for trial participation according to judgment of the Principal Investigator (PI)
* Patients starting afamelanotide 24 hours or more from ictus.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-06-03 (Actual); Primary Completion 2022-02-04 (Actual); Study Completion 2022-02-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Alfred, Melbourne, Australia

REFERENCES:
- [Derived] Stanislaus V, Kam A, Murphy L, Wolgen P, Walker G, Bilbao P, Cloud GC. A feasibility and safety study of afamelanotide in acute stroke patients - an open label, proof of concept, phase iia clinical trial. BMC Neurol. 2023 Jul 26;23(1):281. doi: 10.1186/s12883-023-03338-9. PMID 37496004

RESULTS

PARTICIPANT FLOW:
Groups:
- SCENESSE® (Afamelanotide 16mg): Six adult patients with clots located in the higher segments of the brain and who are ineligible for alternative treatments will be enrolled in the study and evaluated for six weeks. The study will assess patients' brain injury with computed tomography (CT) scans and magnetic resonance imaging (MRI), as well as using recognised methods of clinical evaluation to measure changes in patients' neurological and cognitive function following treatment.
Period: Overall Study
Arm/Group | SCENESSE® (Afamelanotide 16mg)
Started | 6
Completed | 5
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | SCENESSE® (Afamelanotide 16mg)
Number analyzed (Participants) | 6
Age, Continuous [Mean (Full Range); unit: years] | 76.0 [50 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Caucasian | 5
  Race: Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Changes in Volume of Infarct
Time Frame: From Day 0 to Day 3 and Day 0 to Day 9
Measure: Median (Full Range); unit: mL
Arm/Group | SCENESSE® (Afamelanotide 16mg)
Number analyzed (Participants) | 5
mL
  Median change from baseline to Day 3 | 9.97 [1.71 to 59.60]
  Median change from baseline to Day 9 | 4.06 [1.41 to 57.60]
Statistical Analysis 1: Comparison: SCENESSE® (Afamelanotide 16mg); Test type: Other; p = 0.0313, Wilcoxon (Mann-Whitney) — Change from baseline to Day 3
Statistical Analysis 2: Comparison: SCENESSE® (Afamelanotide 16mg); Test type: Other; p = 0.0625, Wilcoxon (Mann-Whitney) — Change from baseline to Day 9

2. Secondary Outcome: Changes of Neurological Function as Measured by the National Institutional Health Stroke Scale (NIHSS).
Description: 0: No stroke symptoms 1-15: Mild to Moderate stroke 16-20: Moderate to severe stroke 21- 42: Severe stroke
Time Frame: From baseline to Day 42
Measure: Median (Full Range); unit: Score on a scale
Arm/Group | SCENESSE® (Afamelanotide 16mg)
Number analyzed (Participants) | 6
Score on a scale | -4.5 [-8 to 41]

3. Secondary Outcome: Changes of Daily Activities as Measured by the Modified Rankin Scale (mRS)
Description: The mRS indicates the degree of disability or dependence in the daily activities of patients who have suffered a stroke or other causes of neurological disability. The scale runs from 0-6, running from perfect health without symptoms (0) to death (+6).
Time Frame: From baseline to Day 42
Measure: Count of Participants; unit: Participants
Arm/Group | SCENESSE® (Afamelanotide 16mg)
Number analyzed (Participants) | 6
Participants
  Pre-stroke score 0 | 4
  Pre-stroke score 1 | 1
  Pre-stroke score 2 | 1
  Day 42 score 3 | 3
  Day 42 score 4 | 2
  Day 42 score 6 | 1

ADVERSE EVENTS:
Time Frame: All adverse events were monitored from baseline until 3 months after the end of treatment, up to 19 weeks.
Description: Patients were advised to report any adverse events to the PI. All adverse events were assessed as unrelated to SCENESSE® (afamelanotide 16 mg).
Arm/Group | SCENESSE® (Afamelanotide 16mg)
All-Cause Mortality (participants affected / at risk) | 1/6
Serious Adverse Events (participants affected / at risk) | 1/6
Other Adverse Events (participants affected / at risk) | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SCENESSE® (Afamelanotide 16mg) (N=6)
Haemorrhagic transformation stroke (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SCENESSE® (Afamelanotide 16mg) (N=6)
Constipation (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Troponin increased (Investigations) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Hypervolaemia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Haemorrhagic transformation stroke (Nervous system disorders) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-04): https://cdn.clinicaltrials.gov/large-docs/03/NCT04962503/Prot_SAP_000.pdf